CLINICAL TRIAL: NCT06585839
Title: Daring Birth - Digital Coaching Solution to Improve Childbirth Experience
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aalto University (Other)
Collaborators: Helsinki University Central Hospital (Other); Business Finland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 6349/2023
Record Dates: First submitted 2024-08-16; First posted 2024-09-19 (Actual); Last update posted 2025-01-31 (Actual); Status verified 2024-09

CONDITIONS: Childbirth Problems; Perinatal Depression; Anxiety in Pregnancy; Pregnancy Related; Postpartum Depression; Postpartum Anxiety; Fear of Childbirth
MeSH Terms: conditions — Depression, Postpartum

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Study (Experimental): Participants have full access to the investigational device, the Natal Mind mobile application.
  Interventions: Behavioral: Digital coaching solution to improve childbirth experience
- Control (Active Comparator): Participants use the investigational device solely for inputting data at predetermined points. They receive standard care without the intervention from the investigational device.
  Interventions: Other: Application for the control group

INTERVENTIONS:
Behavioral: Digital coaching solution to improve childbirth experience — Intervention provides coaching to improve the childbirth experience and offers comprehensive perinatal mental health support to pregnant and postpartum women. It features emotion tracking and exercise customization functionality, along with an avatar-based platform. The app includes digital psychotherapy exercises and psychoeducation. These core elements are complemented by exercises in mindfulness, relaxation, and self-soothing.
  Other Names: Natal Mind
  Arms: Study
Other: Application for the control group — Application for the control group including surveys.
  Arms: Control

SUMMARY:
The aim of the study is to investigate the effectiveness of the Daring Birth digital coaching solution (the Natal Mind app) in enhancing the experience of childbirth. Natal Mind is designed for mobile phones and features a unique blend of emotion tracking, avatar-based interaction, and mass-customized psychoeducation and exercises. These features collectively work to improve the childbirth experience, alleviate pain experience during labor, and mitigate perinatal mental health (PMH) issues namely fear of childbirth (FOC), anxiety, and postpartum depression. The primary outcome of this study is the improvement of the childbirth experience, as it has been recognized to be a fundamental step in preventing postpartum problems.

The study uses a randomized controlled trial (RCT) with two arms: an intervention arm, where participants will have access to the Natal Mind app with its full functionalities, and a control arm, where participants use the app only for answering the study questionnaires while receiving standard care.

ELIGIBILITY:
Inclusion Criteria:

* Nulliparous status Estimated time of delivery (ETD) between 15.5. and 15.9.2024 Between 20 and 28 weeks gestational age at the time of recruitment Fluency in Finnish Intended maternity care and birth hospital located in Finland Aged 18 or above

Exclusion Criteria:

* Referral to a fetal medicine unit Diagnosed psychotic or bipolar disorders Active substance abuse Participation in another clinical study focusing on perinatal mental health

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 200 (Actual)
Dates: Start 2024-02-16 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Childbirth experience Visual Analogue Scale | measured at 3 and 5 weeks postpartum
  Visual Analogue Scale (VAS) for childbirth experience (min 0, max 10; higher scores mean better outcome)
Wijma Delivery Experience Questionnaire | measured at 3 weeks postpartum
  Childbirth experience W-DEQ-B (Wijma Delivery Experience Questionnaire) (min 0, max 165; higher scores mean better outcome)

SECONDARY OUTCOMES:
Fear of childbirth Visual Analogue Scale | measured at baseline, at 30-32 weeks of gestation, and at 35-37 weeks of gestation
  Visual Analogue Scale (VAS) for fear of childbirth (FOC) (min 0, max 10; higher scores mean worse outcome)
Edinburgh Postnatal Depression Scale | measured at 5 weeks postpartum
  Postpartum depression measured with Edinburgh Postnatal Depression Scale (EPDS) (min 0, max 30; higher scores mean worse outcome)
Wijma Delivery Expectancy Questionnaire | measured at 30-32 weeks of gestation
  Fear of childbirth (FOC) measured with Wijma Delivery Expectancy Questionnaire (W-DEQ-A) (min 0, max 165; higher scores mean worse outcome)
Labor pain Visual Analogue Scale | measured at birth and at 5 weeks postpartum
  Visual Analogue Scale (VAS) for labor pain (min 0, max 10; higher scores mean worse outcome)
Generalized Anxiety Disorder | measured at baseline, at 35-37 weeks of gestation, and at 5 weeks postpartum
  Generalized Anxiety Disorder 7-item (GAD-7) (min 0, max 21; higher scores mean worse outcome)

CONTACTS AND LOCATIONS:
Locations (1):
- Aalto University, Espoo, Finland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Related Info — https://daringbirth.com/tutkimus